CLINICAL TRIAL: NCT00165451
Title: Anti-Angiogenic Chemotherapy: A Phase II Trial of Thalidomide, Celecoxib, Etoposide and Cyclophosphamide in Patients With Relapsed or Progressive Cancer
Brief Title: A Trial of Thalidomide, Celecoxib, Etoposide and Cyclophosphamide in Patients With Relapsed or Progressive Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Mark Kieran, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01-046
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Neoplasms
Keywords: Relapsed tumors; Progressive Poor Prognosis Tumors; Thalidomide; Celecoxib; Etoposide; Cyclophosphamide
MeSH Terms: conditions — Neoplasms | interventions — Thalidomide; Celecoxib; Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Thalidomide — Oral administration once daily at night starting at 3mg/Kg for 6 months.
Drug: Celecoxib — Oral administration twice daily starting at 100mg/dose for 6 months.
Drug: Etoposide — Oral administration once daily at night starting at 50mg/m2 3 weeks on and 3 weeks off for 6 months.
  Other Names: VP-16
Drug: Cyclophosphamide — Oral administration once daily at night starting at 3.5mg/m2 3 weeks on and 3 weeks off for 6 months.

SUMMARY:
This study will use a combination of four oral drugs (thalidomide, cyclophosphamide, etoposide and celecoxib) to treat patients with relapsed or progressive cancer. These drugs are expected to target the blood vessels that supply the tumors with what they need to grow.

DETAILED DESCRIPTION:
* Thalidomide will be given orally every evening and the daily dose will escalate until the patient reaches a dose on which they are comfortable and will given continuously for one year.
* Celecoxib will be given orally twice a day and escalated as tolerated for one year.
* Etoposide will be given orally once a day for 21 consecutive days. This medication will alternate with oral cyclophosphamide and will continue for one year.
* Cyclophosphamide will be given orally once a day for 21 consecutive days and as stated above will alternate with etoposide for one year.
* During the treatment, blood tests will be performed every three weeks except during the first 3 week cycle in which testing is performed every 2 weeks. Appropriate imaging studies will be performed every 9 weeks.
* The duration of treatment is one year unless the side effects are too harmful or the tumor grows. Treatment may be continued past one year if the drugs are well tolerated and disease progression has not occured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or progressive poor prognosis tumors for which no curative therapy exists.
* Histologic confirmation of disease at diagnosis or relapse.
* Brain stem glioma patients who have progressed after radiation therapy do not require histologic confirmation. Duration of symptoms at the time of diagnosis must be less than 3 months and should consist of cranial nerve deficits and/or ataxia and/or long tract signs.
* Prior radiation therapy and/or chemotherapy are permitted.
* Karnofsky Performance Status >50. For infants, the Lansky play scale >50% can be substituted.
* Life expectancy > 2 months.
* No active uncontrolled cardiac, hepatic, renal, or psychiatric disease defined as ≥ grade 3 based on the common toxicity criteria.
* No known allergies to sulfonamides
* Adequate renal function: Serum Creatinine < 1.5 mg/dl or creatinine clearance or GFR > 70 ml/min.
* Adequate hepatic function: Total Bilirubin < 1.5 mg/dl; SGOT, SGPT, Alk Phos < 3x normal.(SGOT can be < 4x normal for patients on Zantac).
* Adequate bone marrow reserve: Hgb > 9.0 g/dl, Platelets > 75,000/mm3 (transfusion independent),WBC > 2000/mm3 and ANC > 1000/mm3.
* Patients receiving steroids and/or anti-seizure medications are eligible for this study.

Exclusion Criteria:

* Patients must not be pregnant or nursing, and all patients of child bearing age (both male and female) must be willing to practice birth control during and for 2 months after treatment with thalidomide. If the patient is unable to use oral contraceptives for medical reasons, 2 different barrier methods may be used if approved by the treating physician.
* No concurrent use of other investigational agents.
* Patients that have received more than 2 months of oral therapy with any of the agents used in this study will be ineligible. Standard administration of IV etoposide and cyclophosphamide, usually administered in 3-week cycles is permitted.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2001-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of administering thalidomide, celecoxib, etoposide and cyclophosphamide for recurrent and poor prognosis tumors. | 6 months

SECONDARY OUTCOMES:
To obtain preliminary evidence of biologic activity of these four orally administered | 6 months
to evaluate and document side effects from chronic administration of these four drugs at the doses prescribed in this protocol | 6 months
to evaluate different radiographic techniques as markers of tumor response. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Kieran MW, Turner CD, Rubin JB, Chi SN, Zimmerman MA, Chordas C, Klement G, Laforme A, Gordon A, Thomas A, Neuberg D, Browder T, Folkman J. A feasibility trial of antiangiogenic (metronomic) chemotherapy in pediatric patients with recurrent or progressive cancer. J Pediatr Hematol Oncol. 2005 Nov;27(11):573-81. doi: 10.1097/01.mph.0000183863.10792.d4. PMID 16282886